CLINICAL TRIAL: NCT00870896
Title: The Effects of Tiotropium on the Cough Reflex in Patients With COPD
Brief Title: The Effects of Tiotropium on the Cough Reflex in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ThomasTruncale (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, ThomasTruncale, Associate porfessor, University of South Florida
Organization: University of South Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P65201; 0800000250 V10 (Other Grant/Funding Number: Boehringer Ingelheim)
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
Keywords: capsaicin; COPD; COPD with chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tiotropium (Experimental): Cough reflex measured by capsaicin Inhalation Challenge will follow Dicpinigaitis performed at 1 and 3 months. Solutions prepared to make a stock solution of 0.01 Mol diluted with physiologic saline to yield 11 doubling concentrations from 0.98 to 1,000 uMol/L. Final diluted capsaicin concentrations are: 0.98, 1.95, 3.9, 7.8, 15.6, 31.2, 62.5, 125, 250, 500, and 1000 uMol/L. Then, place 1 ml of the first concentration into nebulizer. Subjects inhale single breath of capsaicin aerosol. Single breaths are delivered in ascending order, with normal saline randomly interspersed to increase blindness, until two or more coughs (C2) and five or more coughs (C5) are reached. The different concentrations are delivered at 2 minute intervals.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — Each subject will then receive Spiriva 18 ug/day for a total of 4 weeks. Each subject will be instructed by the PI on the proper use of the Spiriva inhaler and demonstrate the ability to properly perform the inhalation technique prior to leaving the laboratory. The patient will receive their first dose in the laboratory under the direct supervision of one of the investigators. In addition, subjects will be requested to take their Spiriva inhalation treatment the same time each day.
  Other Names: Spiriva

SUMMARY:
Does tiotropium effect the cough reflex in patients with COPD and chronic bronchitis.

DETAILED DESCRIPTION:
Cough Questionnaire

This questionnaire is designed to assess the impact of cough on various aspects of your life. Read each question carefully and answer by CIRCLING the response that best applies to you. Please answer ALL questions, as honestly as you can.

1. In the last 2 weeks, have you had chest or stomach pains as a result of your cough? 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
2. In the last 2 weeks, have you been bothered by sputum (phlegm) production when you cough? 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
3. In the last 2 weeks, have you been tired because of your cough? 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
4. In the last 2 weeks, have you felt in control of your cough? 1 2 3 4 5 6 7 None of the time Hardly any time A little of the time Some time A good bit of time Most of the time All of the time
5. How often during the last 2 weeks have you felt embarrassed by your coughing? 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
6. In the last 2 weeks, my cough has made me feel anxious 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
7. In the last 2 weeks, my cough has interfered with my job, or other daily tasks 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
8. In the last 2 weeks, I felt that my cough interfered with the overall enjoyment of my life 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
9. In the last 2 weeks, exposure to paints or fumes has made me cough 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time
10. In the last 2 weeks, has your cough disturbed your sleep? 1 2 3 4 5 6 7 All of the time Most of the time A good bit of time Some time A little of the time Hardly any time None of the time

ELIGIBILITY:
Inclusion Criteria:

After signing the informed consent, screening testing will be done to document that a subject meets the requirements of the study. Specific inclusion criteria are:

* Subjects between the ages of 40 and 80 years of age (Dates of Birth 1925-1965)
* Current smoker (with smoking history of > 10 pack/year) or ex-smoker (stopped within 1 year and has at least a 10 pack/year smoking history).
* Subjects will be included if they meet criteria for mild and moderate COPD as defined by the American Thoracic Society and European Respiratory Society position paper. Mild COPD will be defined as a postbronchodilator (2 puffs of albuterol) FEV1/FVC ratio of <0.7 and a predicted FEV1 of > 80%. Moderate COPD will be defined as a postbronchodilator FEV1/FVC ratio of <0.7 and a predicted FEV1 50-80%. A response to bronchodilators is defined as an increase of 12% or 200cc in FEV1 from baseline after inhalation of 2 puffs of albuterol. Both subjects with and without a response to bronchodilators will be included in the study.
* All subjects will be clinically stable for 4 weeks prior to inclusion. Clinical stability is defined as having no recent COPD exacerbations within the last 4 weeks and having received no antibiotics or change in their inhaled steroid dose during that time period. If a subject is on oral steroids, they will be required to be on 10 mg or less each day or no more than 20mg every other day to be eligible. If the oral steroid dose has been titrated over the previous 4 weeks (either up or down) or if the dose is higher than what has been described previously, they will be ineligible for the study.
* All subjects will be off of tiotropium or ipratropium for 1 month prior to the start of the study.
* Chronic cough: Chronic cough will be characterized by the presence of a productive cough for 3 months in each of 2 successive years in persons in whom other causes of chronic cough have been excluded.

Exclusion Criteria:Exclusion Criteria: Subjects will not be eligible for the study if they are

* Age of < 40 or > 80 years.
* Refusal to volunteer for the study and not willing to sign the informed consent form.
* Respiratory disorder other than COPD including asthma, chronic bronchiectasis or pulmonary fibrosis
* Oxygen or ventilator dependent COPD.
* Received any antibiotics or had a change in their inhaled steroid dose during the last 4 weeks. If a subject is on oral steroids, they will be required to be on 10 mg or less each day or no more than 20mg every other day to be eligible. If the oral steroid dose has been titrated over the previous 4 weeks (either up or down) or if the dose is higher than what has been described previously, they will be ineligible for the study.
* History of Congestive heart failure, cardiomyopathy, valvular heart disease, angina, cardiac arrhythmia, or myocardial infarction within the last 6 months or poorly controlled hypertension.
* History of chronic hepatitis or hepatic cirrhosis.
* End-stage renal disease.
* History of neurologic or psychiatric disorder which would interfere with completion of the study.
* Physician diagnosis of Gastroesophageal reflux disease
* Physician diagnosis of allergic, non-allergic rhinitis, or sinusitis
* History of lung cancer
* History of radiation treatment to the chest or mediastinum
* Lung volume reduction surgery, segmentectomy, lobectomy or pneumonectomy
* History of a thoracotomy
* Symptomatic Benign prosthetic hypertrophy
* Symptomatic bladder outlet obstruction
* Symptomatic glaucoma
* Severe COPD defined as a postbronchodilator FEV1/FVC ratio of < 0.7 and a predicted FEV1 of 30-50%. Very severe COPD defined as a postbronchodilator FEV1/FVC ratio of <0.7 and a predicted FEV1 of < 30%. (Eur Respir J 2004; 23: 932-946).
* Within the previous one month (30 days) prior to beginning the study, used or continue to use ipratropium or tiotropium
* Allergic response or history of allergy to lactose

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thoms Truncale, DO,MPH, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - James A Haley Veterans' Hospital, Tampa, Florida
  - University of South Florida (COPH), Tampa, Florida

REFERENCES:
- [Background] Celli BR, MacNee W; ATS/ERS Task Force. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004 Jun;23(6):932-46. doi: 10.1183/09031936.04.00014304. No abstract available. PMID 15219010
- [Background] CIBA Guest symposium Report. Terminology, definitions and classifications of chronic pulmonary emphysema and related conditions. Thorax 1959; 14: 286-289.
- [Background] Standards for the diagnosis and care of patients with chronic obstructive pulmonary disease. American Thoracic Society. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 2):S77-121. No abstract available. PMID 7582322
- [Background] Doherty MJ, Mister R, Pearson MG, Calverley PM. Capsaicin responsiveness and cough in asthma and chronic obstructive pulmonary disease. Thorax. 2000 Aug;55(8):643-9. doi: 10.1136/thorax.55.8.643. PMID 10899239
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Background] Sekizawa K, Jia YX, Ebihara T, Hirose Y, Hirayama Y, Sasaki H. Role of substance P in cough. Pulm Pharmacol. 1996 Oct-Dec;9(5-6):323-8. doi: 10.1006/pulp.1996.0042. PMID 9232670
- [Background] Szallasi A, Blumberg PM. Vanilloid (Capsaicin) receptors and mechanisms. Pharmacol Rev. 1999 Jun;51(2):159-212. No abstract available. PMID 10353985
- [Background] Midgren B, Hansson L, Karlsson JA, Simonsson BG, Persson CG. Capsaicin-induced cough in humans. Am Rev Respir Dis. 1992 Aug;146(2):347-51. doi: 10.1164/ajrccm/146.2.347. PMID 1489123
- [Background] Fujimura M, Sakamoto S, Kamio Y, Matsuda T. Effects of methacholine induced bronchoconstriction and procaterol induced bronchodilation on cough receptor sensitivity to inhaled capsaicin and tartaric acid. Thorax. 1992 Jun;47(6):441-5. doi: 10.1136/thx.47.6.441. PMID 1386691
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10/14/08 to 2/5/09
Pre-assignment Details: Unable to recruit 20 participates study stopped at 5
Groups:
- Group 1: Capsaicin Inhalation challenge (CIH): Each solution of capsaicin administered to a subject will be quantified by HPLC. Solutions of capsaicin are prepared to make a stock solution of 0.01 Mol and subsequently further diluted with physiologic saline solution to yield 11 serial doubling concentrations from 0.98 to 1,000 uMol/L. Final diluted capsaicin concentrations are: 0.98, 1.95, 3.9, 7.8, 15.6, 31.2, 62.5, 125, 250, 500, and 1000 uMol/L. Single breaths of capsaicin are delivered in ascending order, with normal saline solution randomly interspersed to increase challenge blindness, until two or more coughs (C2) and five or more coughs (C5) are reached. The different concentrations are delivered at 2 minute intervals. CIH is administered at baseline one and 3 months following treatment with Spiriva
Period: Overall Study
Arm/Group | Group 1
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty male subjects between 40-80 years of age with COPD will be recruited from the USF and James A. Haley medical clinics, word of mouth, newspaper and radio advertising. We are restricting the study to men because woman have a more sensitive cough reflex and analysis of data will be more difficult when comparing as a group.
Groups:
- Tiotropium: Subjects 40-80 with > 10 pk/year or ex-smoker stopped within 1 year with 10 pk/year smoking history, Subjects with mild and moderate COPD defined by ATS/ERS clinically stable for 4 weeks, subjects off tiotropium or ipratropium 1 month prior to start, Chronic cough Defined by ATS/ERS Exclusion:Age < 40 or > 80, Refusal to volunteer, Lung disease other than COPD,O2 or ventilator dependent COPD, Received antibiotics or a change in inhaled steroid during last 4 weeks.History CHF, cardiomyopathy, valvular heart disease, angina, arrhythmia, MI or uncontrolled HTN within last 6 months, History chronic hepatitis/cirrhosis, End-stage renal disease, neurologic or psychiatric disorder, Physician diagnosis GERD/allergic/non-allergic rhinitis/sinusitis/lung cancer/radiation to the chest or mediastinum/Lung volume reduction surgery/lobectomy/pneumonectomy/thoracotomy, Symptomatic BPH/bladder outlet obstruction/glaucoma Severe COPD defined ERS/ATS, Allergic response or history of allergy to lactose
Arm/Group | Tiotropium
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Coughs Following Capsaicin Inhalation Challenge at Baseline and Following 30 Days of Treatment With Spiriva (Baseline and 30 Days)
Description: We measured the change in the number of coughs following capsaicin inhalation challenge from baseline followed by 30 days of treatment with spiriva
Time Frame: 30 days
Population: Power two-sided t-test for C5. our previous studies coefficient of variation for C5 was 3.2%. We propose power 0.80/significance 0.05. multiple comparisons utilize Bonferroni procedure significance will be 0.017 ability to detect minimum difference of 3.7 uMol. Thus, if alpha 0.05 and beta 0.20, to detect difference require 20 subjects each group.
Measure: Mean (Standard Deviation); unit: coughs per dose of capsaicin
Groups:
- Group 1: Capsaicin Inhalation Challenge Testing (CICT) will follow the protocol of Dicpinigaitis et al (Chest 2003; 123:685-8). CICT will be performed at baseline before beginning treatment with tiotropium and at 4 weeks after initiation of treatment. Solutions of capsaicin are prepared to make a stock solution of 0.01 Mol and subsequently further diluted with physiologic saline solution to yield 11 serial doubling concentrations from 0.98 to 1,000 uMol/L. Final diluted capsaicin concentrations are: 0.98, 1.95, 3.9, 7.8, 15.6, 31.2, 62.5, 125, 250, 500, and 1000 uMol/L. Single breaths of capsaicin are delivered in ascending order, with normal saline solution randomly interspersed to increase challenge blindness, until five or more coughs (C5) are reached. We measured the change in the number of coughs at baseline and following 30 days of treatment with spiriva
Arm/Group | Group 1
Number analyzed (Participants) | 5
coughs per dose of capsaicin | 2.5 (2.75)

2. Secondary Outcome: Change in FEV1 (in Liters)
Description: Change in FEV1 ( in liters) at baseline and following 30 days of treatment with Spiriva
Time Frame: 30 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters
Groups:
- Spirometry: We measured the change in FEV1 (in liters) at baseline and following 30 days of treatment with Spiriva.Spirometry will be performed with a KoKO Spirometer, which uses a pneumotachograph to provide Flow/Volume Loops and Volume/Time graphics and multiple incentive graphics for patient coaching. Spirometry will be performed at baseline and at 4 weeks. Normal values will be those of Hankinson, et al (Am J Respir Crit Care Med 159:179-187). Spirometry will also be performed after each dose of inhaled capsaicin. If there is a drop of 20% or more in FEV1 at any time after inhalation of capsaicin, the protocol will be ended at that point.
Arm/Group | Spirometry
Number analyzed (Participants) | 5
liters | .315 (138)

3. Secondary Outcome: Change in FEV1/FVC Ratio
Description: We measured the change in FEV1/FVC ratio at baseline and following 30 days of treatment with Spiriva.Change in ratio reflects the percentage value (ratio) at 30 days minus the percentage value (ratio) at baseline x 100
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Change in FEV1/FVC: We measured the change in FEV1/FVC ratio before and after treatment with Spiriva. Change in ratio reflects the percentage value at 30 days minus the percentage value at baseline
Arm/Group | Change in FEV1/FVC
Number analyzed (Participants) | 5
percentage change | 3 (5.74)

ADVERSE EVENTS:
Arm/Group | Tiotropium
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes